CLINICAL TRIAL: NCT01445288
Title: An Exploratory Study of Biologic and Pathophysiologic Effects of Radiation Therapy in Pediatric Patients With Central Nervous System Tumors
Brief Title: Exploratory Study of Effects of Radiation Therapy in Pediatric Patients With Central Nervous System Tumors
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060219; 06-C-0219
Record Dates: First submitted 2011-09-30; First posted 2011-10-03 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-10-24

CONDITIONS: Diffuse Intrinsic Pontine Glioma; PNET; Ependymoma; Germinoma; Medulloblastoma
Keywords: Neurotoxicity; Brain Tumor; Children; Angiogenesis; Imaging; Natural History; Central Nervous System Tumor; CNS Tumor
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma; Neuroectodermal Tumors, Primitive; Ependymoma; Germinoma; Medulloblastoma; Neurotoxicity Syndromes; Brain Neoplasms; Central Nervous System Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Pediatric Patients with Central Nervous System Tumors

SUMMARY:
This study will analyze the effects of radiation given to children who have tumors of the central nervous system (CNS). Researchers want to learn more about changes in the quality of life that patients may experience as a result of radiation.

Patients ages 21 and younger who have a primary CNS tumor and who have not received radiation previously may be eligible for this study. They will have a medical history and physical examination. Collection of blood (about 2-1/2 tablespoons) and urine will be done, as well as a pregnancy test. Patients will complete neuropsychological tests, which provide information about their changes in functioning over time. An expert in psychology will give a number of tests, and the patient's parents or guardian will be asked to complete a questionnaire about the patient's behavior. Also, patients will be given a quality of life questionnaire to complete and vision and hearing tests. The radiation itself is prescribed by patients' doctors and is not part of this study.

Magnetic resonance imaging (MRI) will give researchers information about the tumor and brain, through several scanning sequences . MRI uses a strong magnetic field and radio waves to obtain images of body organs and tissues. Patients will lie on a table that slides into the enclosed tunnel of the scanner. They will need to lie still, and medication may be given to help them to do that. They may be in the scanner for up to 2 hours. As the scanner takes pictures, patients will hear knocking or beeping sounds, and they will wear earplugs to reduce the noise. A contrast agent will be administered, to allow images be seen more clearly. Blood and urine tests will be conducted after the first dose of radiation. MRI scans will be done 2 weeks after patients finish radiation therapy and again at 6 to 8 weeks, 6 months, 12 months, and yearly. Also at those follow-up periods, patients will undergo similar procedures as previously, including blood and urine tests and neuropsychological testing. Patients can remain in this study for 5 years.

DETAILED DESCRIPTION:
Background:

This exploratory study will be performed in pediatric patients with CNS tumors who are undergoing radiation therapy to investigate pathophysiologic effects of radiation on the CNS. The study includes the analysis of blood, urine, and CSF (if available) to measure biological markers involved with angiogenesis, blood: brain barrier integrity, and neurotoxicity. It also entails comprehensive MR imaging techniques and neuropsychological testing in an effort to correlate changes with biomarker measurements.

Objectives:

1. To detect changes in angiogenesis related to radiation of the CNS by:

   * Measurement of VEGF, bFGF, thrombospondin, TNF-alpha, IL-12, IL-8, and MMP in blood and urine specimens.
   * MR perfusion and DEMRI.
2. To describe changes in blood:brain barrier permeability associated with radiation of the CNS.
3. To characterize neurotoxicity by:

   * Measuring biomarkers associated with neurotoxicity
   * Documenting changes in neurobehavioral functioning through longitudinal comprehensive assessments
   * Describing changes in quality of life (QOL)
   * Assessing changes in memory
   * Defining changes in ophthalmologic studies associated with radiation.
   * Detecting changes in audiometry associated with radiation.

Eligibility Criteria:

* Patients must have a primary CNS tumor for which radiation therapy is recommended.
* Patients must be less than or equal to 21 years of age.
* Prior/Concurrent: Patients will be eligible if they have not received prior radiation. Patients who have undergone surgery or received chemotherapy are eligible.
* Performance Status: Patients will be eligible regardless of performance score.

Design:

This minimally invasive study is designed to explore various biologic effects of radiation on the pediatric CNS in an attempt to 1) obtain information on the pathophysiology of radiation-induced damage, 2) explore the association of neuropsychological deficits with biologic markers and neuroimaging abnormalities, 3) document changes in neurobehavioral functioning through longitudinal comprehensive neuropsychological assessments with comparison of various radiation therapy techniques, 4) describe changes in quality of life in pediatric patients who have received radiation therapy, and 5) attempt to identify children at increased risk of radiation-induced neurotoxicity.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age: Patients must be less than or equal 21 years of age.

Tumor: Any primary CNS tumor.

Referred for radiation therapy at NCI.

Signed informed consent by patient, parent or legal guardian.

PERFORMANCE SCORE: any.

PRIOR/CONCURRENT THERAPY: Patients will be eligible if they have not received prior radiation.

Patients who have undergone prior surgery or who have received chemotherapeutic regimens are eligible.

EXCLUSION CRITERIA:

Patients who have received prior radiation.

Patients who are unable to have MRI performed for any reason.

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients 21 years of age or younger with CNS tumors for which radiation therapy is recommended@@@
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2006-12-05 (Actual)

PRIMARY OUTCOMES:
Measure changes in antiogenesis, blood brain barrier permability and neurotoxicity re to radiation of the CNS | before and up to 8 years after
  Measurement of VEGF, bFGF, thrombospondin, TNF-a, IL-12, IL-8, and MMP in blood and urine specimens

SECONDARY OUTCOMES:
Describe changes in imaging, endocrine function after xrt to the brain | before and up to 8 years after
  Measurement of S100-beta and transthyretin in blood
Monitor changes in serum proteome and germline polymorphisms | before and up to 8 years after
  Assesed changed in memory, QOL, neurobehavioral functioning, ophthalmologic studies, and audiometry associated with radiation

CONTACTS AND LOCATIONS:
Overall Officials: John W Glod, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as the database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Background] Garcia-Barros M, Paris F, Cordon-Cardo C, Lyden D, Rafii S, Haimovitz-Friedman A, Fuks Z, Kolesnick R. Tumor response to radiotherapy regulated by endothelial cell apoptosis. Science. 2003 May 16;300(5622):1155-9. doi: 10.1126/science.1082504. PMID 12750523
- [Background] Wyllie AH, Kerr JF, Currie AR. Cell death: the significance of apoptosis. Int Rev Cytol. 1980;68:251-306. doi: 10.1016/s0074-7696(08)62312-8. No abstract available. PMID 7014501
- [Background] Mulhern RK, Hancock J, Fairclough D, Kun L. Neuropsychological status of children treated for brain tumors: a critical review and integrative analysis. Med Pediatr Oncol. 1992;20(3):181-91. doi: 10.1002/mpo.2950200302. PMID 1574027
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2006-C-0219.html